CLINICAL TRIAL: NCT05936333
Title: Exploration of Allograft Humoral Rejection in Chronic Histiocytic Intervillositis
Acronym: RH-PL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: APHP221169
Record Dates: First submitted 2023-06-12; First posted 2023-07-07 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-10

CONDITIONS: Chronic Histiocytic Intervillositis; Intrauterine Growth Retardation; Fetal Death in Utero; Miscarriage
MeSH Terms: conditions — Fetal Growth Retardation; Stillbirth; Abortion, Spontaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patient with chronic histiocytic intervillositis (Experimental): Patient with CHI, as well as her children and their father. Blood collection from the parents, saliva collection (or blood collection) from the children, placenta collection
  Interventions: Procedure: Biological collection
- patients with anti-phospholipid syndromes (APS) (Active Comparator): Patient with antiphospholipid syndrome, as well as her children and their father. Blood collection from the parents, saliva collection (or blood collection) from the children, placenta collection
  Interventions: Procedure: Biological collection
- women with a third full-term pregnancy without growth retardation. (Placebo Comparator): Patient with normal pregnancies, as well as her children and their father. Blood collection from the parents, saliva collection (or blood collection) from the children, placenta collection
  Interventions: Procedure: Biological collection

INTERVENTIONS:
Procedure: Biological collection — up to 25 mL of blood collection for the adults and saliva collection for the minor at inclusion, and placenta collection at childbirth

SUMMARY:
Chronic histiocytic intervillositis (CHI) is a rare condition with an incidence of 5 in 10,000 pregnancies. This rare condition is associated with placental inflammatory lesions leading to severe and recurrent obstetrical complications: intrauterine growth retardation (IUGR), fetal death in utero and miscarriage. The pathophysiological mechanisms of CHI are poorly understood, while the empirical treatments prescribed to prevent recurrence are cumbersome and of poor efficacy.

Recent findings suggest that an alloimmune response may play a role. In a recent work, the investigators have demonstrated the role of maternal alloantibodies directed against fetal HLA antigens in two patients followed for recurrent IUGR associated with CHI. Their work suggests that a humoral alloimmune response directed against fetal HLA antigens mimics an allograft rejection process.

The investigators propose to extend the preliminary results obtained in these patients to provide new insights into the pathophysiological mechanisms of CHI, and eventually to predict the risks of fetal loss.

ELIGIBILITY:
Family Inclusion Criteria:

* Mother and father ≥ 18 years old
* For mothers in the CHI group :

  * History of a normal pregnancy (full term, alive child) or IUGR/MFIU or miscarriage(s) or abortion followed by at least 1 obstetrical complication such as IUGR, MFIU, miscarriage
  * Diagnosis of chronic histiocytic intervillitis made by placental anatomopathological examination with CD68+ marking
* For the mothers of the antiphospholipid syndrom group

  * History of miscarriage(s)
  * Having an anti-phospholipid syndrome
* For mothers in the normal pregnancy group:

  * Third consecutive pregnancy of normal course, at term (≥ 36 weeks of amenorrhea) with eutrophic child

For the mother and father:

o Consent to participate in the study and for the participation in the study of at least one child and/or the use of existing samples (placenta / fetal DNA) from at least one previous pregnancy with CHI for the CHI group or at least one previous miscarriage for the APS group

For the father:

o Father of the last pregnancy and of the child(ren) participating in the study

Exlusion criteria :

* For mothers in the normal pregnancy group:

  o Suspected or confirmed intra-amniotic infection
* For all the mothers:

  * History of blood transfusion
  * History of allogeneic organ transplantation
* For the mother and the father:

  * Person under legal protection (guardianship, curatorship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-10-11 (Actual); Primary Completion 2025-10-11 (Estimated); Study Completion 2025-10-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients diagnosed with CHI, defined by the concomitant presence of the 3 criteria required to evoke humoral alloimmune rejection for this pathology | up to 6 months
  Proportion of patients diagnosed with CHI, defined by the concomitant presence of the 3 criteria required to evoke humoral alloimmune rejection for this pathology, namely CD68+ infiltrate, AND C4d deposits on the trophoblastic villi AND the presence of at least one FSA (fetus-specific antibody, directed against fetal HLA antigens in the maternal blood) with an elevated level, defined by a Mean Fluorescence Intensity (MFI) > 10,000).
  This proportion of patients observed in CHI carriers will be compared to the proportion of patients with the concomitant presence of the same 3 criteria observed in the other two control groups.

SECONDARY OUTCOMES:
To measure the FSA levels by Mean Fluorescence Intensity for the different obstetrical complications: intrauterine growth retardation (IUGR), fetal death in utero and abortion for IUGR. | up to 6 months
to measure the correlation between fetus-specific antibody level by Mean Fluorescence Intensity and the severity and/or precocity of obstetrical complications | up to 6 months
measure of semi-quantitative graduation of C4d in placenta compared to percentage of villositis | up to 6 months
measure of semi-quantitative graduation of CD68+ infiltrate in placenta compared to surface and number of involved villositis | up to 6 months
To measure the expression of HLA class I and II molecules by placental villi by ß2-microglobulin and HLA-DR labelling | up to 6 months
Epitope analysis with algorithm developped by laboratoire HLA de St Louis (Pr JL Taupin) | up to 6 months
  Epitope analysis with algorithm developped by laboratoire HLA de St Louis (Pr JL Taupin) to determine whether an antibody response against a limited number of epitopes present during a first pregnancy that resulted in a healthy child can explain immunization against both paternal alleles

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra LETOURNEAU, Doctor, Principal Investigator — APHP, Antoine Béclère Hospital, CLAMART, France
Locations (1):
- Antoine Béclère Hospital, Clamart, France

IPD SHARING:
Plan to Share IPD: No